CLINICAL TRIAL: NCT05868941
Title: Efficacy and Safety of Broncho Muco Cleaner Balloon Dilation Therapy in Chronic Bronchitis-predominant COPD Cases
Brief Title: Efficacy and Safety of Broncho Muco Cleaner Balloon Dilation Therapy
Acronym: EXERTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinodevice (Industry)
Collaborators: Klinar CRO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K-BB001-EXERTION
Record Dates: First submitted 2022-02-24; First posted 2023-05-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: COPD
Keywords: Chronic Bronchitis; Medical Device; Baloon Dilatation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, prospective local medical device clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Broncho Muco Cleaner (Experimental): It will be applied to patients with a diagnosis of chronic bronchitis-predominant COPD, who cannot achieve adequate clinical and functional improvement despite optimal medical therapy. In patients who meet the patient selection criteria, anesthesia approval will be obtained before the procedure will be performed under general anesthesia
  Interventions: Device: Broncho Muco Cleaner

INTERVENTIONS:
Device: Broncho Muco Cleaner — The endotracheal tube will be passed with a bronchoscope. During the procedure, the product is connected to the oxygen jack in the hospital, inflated and deflated, turning the thickened goblet cell layer that causes sputum production to foamy liquid. For the procedure, it will be entered through the intubation tube with a fiberoptic bronchoscope, and the airways with a diameter of 3 to 8 mm, primarily the airways, and all the respiratory tract mucosa that can be reached will be treated with a balloon in a total of 3 sessions. For these procedures, balloons selected in accordance with the diameter of the bronchi will be used in the respiratory tract.
  In patients who meet the patient selection criteria, intervention will be made with a balloon that inflates and deflates at the determined frequency and pressure from the subsegment level that can be reached with the bronchoscope to the inner surface of the airways proximally.

SUMMARY:
In COPD patients with chronic bronchitis, it is aimed to determine whether the broncho muco cleaner balloon dilation method can provide clinical and functional benefit by causing destruction in hyperplasic goblet cells in the bronchial system. Although 2 studies have been published on this subject before, one of them is a retrospective design and the other is a pilot study consisting of only 10 patients . Therefore, it is clear that it should be supported by a controlled prospective study with more patients.

Within the scope of the research, broncho muco cleaner balloon dilatation treatment will be performed with fiberoptic bronchoscope under general anesthesia in chronic bronchitis-predominant COPD cases, and the effectiveness and reliability of the procedure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes aged 40-75 years
* Being diagnosed with stage II-IV chronic bronchitis-predominant COPD according to the GOLD guideline
* To have quit smoking for at least 6 months
* mMRC 2 and above
* Receiving optimal medical treatment for COPD
* Being stable for at least 3 weeks
* To have completed 6 weeks of pulmonary rehabilitation before the first procedure
* Having sufficient mental and physical capacity to sign the voluntary consent form for the procedure.

Exclusion Criteria:

* be under the age of 40 and over the age of 75
* pregnant patients
* breastfeeding a child
* Being an active smoker
* Concurrent asthma
* Chronic kidney disease with GFR <30 ml/min
* Clinically significant arrhythmia, Left heart failure (EF<45) or pulmonary hypertension (PABs>45 mmHg)
* Liver cirrhosis
* Those who use anticoagulants or clopidogrel or equivalent drugs and cannot be stopped before and during the procedure, or the presence of bleeding diathesis
* 6 minutes walking test <100 meters
* FEV1<15%
* Those with positive early reversibility in pulmonary function tests
* Patients who do not regularly take 15lgu15in therapy for COPD
* Emphysema-predominant COPD patients
* Presence of active malignancy
* Partial CO2 pressure > 55mmHg or pO2<55 mmHg in room air
* Active pulmonary infection
* Pneumothorax or pulmonary surgery in the last 6 months
* Patients with other clinically significant lung disease other than COPD
* Those who have undergone a previous lung device procedure, including implanted emphysema stents, lung coil delivery, valves, lung denervation, or other devices for emphysema.
* Those taking > 10 mg of prednisolone per day
* Those with a known sensitivity to the drug (such as lidocaine, 15lgu15ine and benzodiazepines) needed to perform bronchoscopy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Reliability of the procedure - Safety | 52 weeks
  Reliability of the procedure (adverse events occurring) for 52 weeks post-procedure.
Patients' Tolerence - mMRC dyspnea scale | 52 Weeks
  Within the scope of the KBB001 Exertion Study, the broncho muco cleaner procedure to be applied to the patients will be performed with fiberoptic bronchoscopy under general anesthesia. Any undesirable event that may be associated with and after the transaction will be recorded. Primary evaluation criteria in determining the Processing efficiency of your device.
Patients' Tolerence - COPD Exacerbation Number (severity of exacerbation will be indicated as mild, moderate, severe.) | 52 Weeks
  Within the scope of the KBB001 Exertion Study, the broncho muco cleaner procedure to be applied to the patients will be performed with fiberoptic bronchoscopy under general anesthesia. Any undesirable event that may be associated with and after the transaction will be recorded. primary evaluation criteria in determining the Processing efficiency of your device
Patients' Tolerence - St George Respiratory Questionnaire | 52 Weeks
  Within the scope of the KBB001 Exertion Study, the broncho muco cleaner procedure to be applied to the patients will be performed with fiberoptic bronchoscopy under general anesthesia. Any undesirable event that may be associated with and after the transaction will be recorded. primary evaluation criteria in determining the Processing efficiency of your device.
Patients' Tolerence - 6 min walking test | 52 Weeks
  Within the scope of the KBB001 Exertion Study, the broncho muco cleaner procedure to be applied to the patients will be performed with fiberoptic bronchoscopy under general anesthesia. Any undesirable event that may be associated with and after the transaction will be recorded. primary evaluation criteria in determining the Processing efficiency of your device.
Patients' Tolerence - Pulmonary Function Test (FEV1, FVC values in (lt) and (%) values as well as FEV1/ FVC rate (in %) | 52 Weeks
  Within the scope of the KBB001 Exertion Study, the broncho muco cleaner procedure to be applied to the patients will be performed with fiberoptic bronchoscopy under general anesthesia. Any undesirable event that may be associated with and after the transaction will be recorded. primary evaluation criteria in determining the Processing efficiency of your device.
Detection of Execerbations | 52 weeks
  COPD Exacerbation (COPD Exacerbation) is one of the most important problems of COPD patients and includes the risk of mortality and mirdit. It is expected that the number of exacerbations of the patients will decrease with the broncho muco cleaner balloon treatment. The number and severity of exacerbations (mild, moderate, severe) at each visit of the patient will be noted to assess the effect of treatment on exacerbations.
Quality of Life for the device | 52 Weeks
  A St George quality of life survey will be conducted and recorded. Every 4-point change in the SGRQ questionnaire will be considered minimal clinical significance.

SECONDARY OUTCOMES:
Improvement in functional parameters - 6 Minute Walk Test (V1-V6) | 52 weeks
  - 6 Minute Walk Test (V1-V6)
Improvement in functional parameters - Pulmonary Function Test (V1-V2-V3-V4-V5-V6) | 52 weeks
  - Pulmonary Function Test (V1-V2-V3-V4-V5-V6)
Adverse events | 52 weeks
  Adverse events seen (AE)
Changes in laboratory test results | 52 weeks
  Change in blood chemistry tests and hemogramcompared to baseline and EoT

CONTACTS AND LOCATIONS:
Overall Officials: Erdogan Cetinkaya, Principal Investigator — stanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital
Locations (1):
- Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided